CLINICAL TRIAL: NCT00398840
Title: A Phase 1 Dose Escalation Study of ARQ 171 in Adult Patients With Advanced Solid Tumors
Brief Title: A Study of ARQ 171 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Arqule, Arqule, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 171-101
Record Dates: First submitted 2006-11-09; First posted 2006-11-14 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Cancer
Keywords: Cancer; Solid Tumors; advanced solid tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ARQ 171

SUMMARY:
This is an open label, dose escalation study of ARQ 171 administered via intravenous infusion (IVI) into a peripheral vein weekly.

Patients with advanced solid tumors, who are refractory to available therapy or for whom no standard systemic therapy exists, will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be obtained and documented prior to study-specific screening procedures.
* A histologically or cytologically confirmed advanced solid tumor
* ≥ 18 years of age
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors
* Karnofsky performance status ≥ 70%
* Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after participation.
* Females of childbearing potential must have a negative serum pregnancy test.
* Laboratory results must meet study criteria.

Exclusion Criteria:

* Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within four weeks of first infusion
* Surgery within 4 weeks prior to first infusion
* Known untreated brain metastases
* Pregnant or breastfeeding
* Uncontrolled intercurrent illness, or uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements
* Other cancer within the last five years, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri or basal or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability and maximum tolerated dose (MTD) of ARQ 171

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile of ARQ 171
To assess the preliminary anti-tumor activity of ARQ 171

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Premiere Oncology, Santa Monica, California
  - Dana Farber/Harvard Cancer Center, Boston, Massachusetts
  - Mary Crowley Medical Research Center, Dallas, Texas